CLINICAL TRIAL: NCT01114217
Title: A Phase III, Open-Label Extension Trial of the Safety and Efficacy of Ferumoxytol for the Episodic Treatment of Iron Deficiency Anemia
Brief Title: A Trial of Ferumoxytol for the Episodic Treatment of Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-FER-IDA-303
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia; Feraheme; Ferumoxytol; IDA
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ferumoxytol (Experimental): Participants received ferumoxytol or placebo during AMAG-FER-IDA-301 [NCT01114139]. Participants enrolled in AMAG-FER-IDA-303, a 6-month Extension Study, were evaluated monthly and could receive treatment with ferumoxytol only if they met criteria defined as persistent or recurrent IDA, hemoglobin <11.0 grams per deciliter (g/dL) and transferrin saturation (TSAT) <20% at any evaluation visit, (except study termination visit). Participants who met criteria began a 5-week treatment period (TP) and received 2 doses of ferumoxytol 510 mg intravenously (IV). The first IV 510-mg dose was administered on TP Day 1 (Baseline); the second 2-8 (5±3) days after Dose 1. The first treatment course with ferumoxytol for participants who previously received placebo in AMAG-FER-IDA-301 was considered Course 1; Course 2 included participants who previously received ferumoxytol in AMAG-FER-IDA-301; subsequent treatment courses were serially numbered.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — IV Ferumoxytol
  Other Names: Feraheme

SUMMARY:
To evaluate the safety and efficacy of ferumoxytol for the episodic treatment of iron deficiency anemia (IDA).

ELIGIBILITY:
Key Inclusion Criteria include:

1. Participants who completed participation in study AMAG-FER-IDA-301 [NCT01114139]
2. Female participants of childbearing potential who are sexually active must be on an effective method of birth control and agree to remain on birth control until completion of participation in the study

Key Exclusion Criteria include:

1. Experienced a serious adverse event (SAE) related to ferumoxytol in study AMAG-FER-IDA-301
2. Female participants who are pregnant, intend to become pregnant, are breastfeeding, or have a positive serum/urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2010-07-27 (Actual); Primary Completion 2012-09-24 (Actual); Study Completion 2013-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (79):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, Mobile, Alabama
  - Clinical Trial Site, Montgomery, Alabama
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Anaheim, California
  - Clinical Trial Site, Bakersfield, California
  - Clinical Trial Site, Buena Park, California
  - Clinical Trial Site, Colton, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Mission Hills, California
  - Clinical Trial Site, Orange, California
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Pueblo, Colorado
  - Clinical Trial Site, Bristol, Connecticut
  - Clinical Trial Site, Groton, Connecticut
  - Clinical Trial Site, Boynton Beach, Florida
  - Clinical Trial Site, Clearwater, Florida
  - Clinical Trial Site, Hialeah, Florida
  - Clinical Trial Site, Holiday, Florida
  - Clinical Trial Site, Inverness, Florida
  - Clinical Trial Site, Margate, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Miami Lakes, Florida
  - Clinical Trial Site, Naples, Florida
  - Clinical Trial Site, Vero Beach, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Zephyrhills, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Decatur, Georgia
  - Clinical Trial Site, Dublin, Georgia
  - Clinical Trial Site, Sandy Springs, Georgia
  - Clinical Trial Site, Stockbridge, Georgia
  - Clinical Trial Site, Aurora, Illinois
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Skokie, Illinois
  - Clinical Trial Site, Springfield, Illinois
  - Clinical Trial Site, Wichita, Kansas
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Bethesda, Maryland
  - Clinical Trial Site, Hollywood, Maryland
  - Clinical Trial Site, Bay City, Michigan
  - Clinical Trial Site, Wyoming, Michigan
  - Clinical Trial Site, Kansas City, Missouri
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, Lawrenceville, New Jersey
  - Clinical Trial Site, Neptune City, New Jersey
  - Clinical Trial Site, Plainsboro, New Jersey
  - Clinical Trial Site, Voorhees Township, New Jersey
  - Clinical Trial Site, Albuquerque, New Mexico
  - Clinical Trial Site, Brooklyn, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Raleigh, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Canton, Ohio
  - Clinical Trial Site, Carlisle, Ohio
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Marion, Ohio
  - Clinical Trial Site, Mentor, Ohio
  - Clinical Trial Site, Middletown, Ohio
  - Clinical Trial Site, Zanesville, Ohio
  - Clinical Trial Site, Norman, Oklahoma
  - Clinical Trial Site, Jenkintown, Pennsylvania
  - Clinical Trial Site, Levittown, Pennsylvania
  - Clinical Trial Site, Columbia, South Carolina
  - Clinical Trial Site, Greer, South Carolina
  - Clinical Trial Site, Myrtle Beach, South Carolina
  - Clinical Trial Site, North Charleston, South Carolina
  - Clinical Trial Site, Rapid City, South Dakota
  - Clinical Trial Site, Arlington, Texas
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Laredo, Texas
  - Clinical Trial Site, Longview, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Orem, Utah
  - Clinical Trial Site, Chesapeake, Virginia
  - Clinical Trial Site, Norfolk, Virginia
- Canada (6):
  - Clinical Trial Site, Vancouver, British Columbia
  - Clinical Trial Site, Saint John, New Brunswick
  - Clinical Trial Site, London, Ontario
  - Clinical Trial Site, Thornhill, Ontario
  - Clinical Trial Site, Vaughan, Ontario
  - Clinical Trial Site, Pointe-Claire, Quebec
- Hungary (5):
  - Clinical Trial Site, Békéscsaba
  - Clinical Trial Site, Gyula
  - Clinical Trial Site, Komárom
  - Clinical Trial Site, Szekszárd
  - Clinical Trial Site, Vác
- India (12):
  - Clinical Trial Site, Hyderabad, Andhra Pradesh
  - Clinical Trial Site, Secunderabad, Andhra Pradesh
  - Clinical Trial Site, Guwahati, Assam
  - Clinical Trial Site, Bangalore, Karnataka
  - Clinical Trial Site, Aurangabad, Maharashtra
  - Clinical Trial Site, Nagpur, Maharashtra
  - Clinical Trial Site, Nashik, Maharashtra
  - Clinical Trial Site, Pune, Maharashtra
  - Clinical Trial Site, Jaipur, Rajasthan
  - Clinical Trial Site, Chennai, Tamil Nadu
  - Clinical Trial Site, Madurai, Tamil Nadu
  - Clinical Trial Site, Lucknow, Uttar Pradesh
- Latvia (4):
  - Clinical Trial Site, Daugavpils
  - Clinical Trial Site, Riga
  - Clinical Trial Site, Valmiera
  - Clinical Trial Site, Ventspils
- Poland (4):
  - Clinical Trial Site, Bialystok
  - Clinical Trial Site, Sopot
  - Clinical Trial Site, Warsaw
  - Clinical Trial Site, Wroclaw

REFERENCES:
- [Background] Vadhan-Raj S, Ford DC, Dahl NV, Bernard K, Li Z, Allen LF, Strauss WE. Safety and efficacy of ferumoxytol for the episodic treatment of iron deficiency anemia in patients with a history of unsatisfactory oral iron therapy: Results of a phase III, open-label, 6-month extension study. Am J Hematol. 2016 Feb;91(2):E3-5. doi: 10.1002/ajh.24240. No abstract available. PMID 26572233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who previously enrolled in and completed AMAG-FER-IDA-301 [NCT01114139], received any dose of study drug, and met the inclusion/exclusion criteria were eligible to enroll in this Extension Study AMAG-FER-IDA-303.
Groups:
- Received Ferumoxytol in IDA-303: Participants received ferumoxytol or placebo during AMAG-FER-IDA-301 [NCT01114139]. Participants enrolled in AMAG-FER-IDA-303 who were found to have persistent or recurrent iron deficiency anemia (IDA), defined as hemoglobin <11.0 grams per deciliter (g/dL) and transferrin saturation (TSAT) <20% at any monthly evaluation visit (with the exception of the Study Termination visit), began a 5-week Treatment Period (TP) and received a total of 2 doses of ferumoxytol 510 milligrams (mg) intravenously (IV). The first IV 510 mg dose was administered on TP Day 1 (baseline) and second dose 2 to 8 (5±3) days after Dose 1, for a total cumulative dose of 1.02 grams (g).
- Did Not Receive Ferumoxytol in IDA-303: Participants who received ferumoxytol or placebo during AMAG-FER-IDA-301 [NCT01114139] and did not receive ferumoxytol during AMAG-FER-IDA-303.
Period: Overall Study
Arm/Group | Received Ferumoxytol in IDA-303 | Did Not Receive Ferumoxytol in IDA-303
Started | 337 | 297
Received at Least 1 Dose of Ferumoxytol | 337 | 0
Completed (Completed Study is defined as had study drug and Week 5 visit.) | 262 (Two participants lacked study completion data: one site stopped communicating during the study.) | 199
Not Completed | 75 | 98
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 17 | 33
Not completed — Withdrawal by Subject | 21 | 28
Not completed — Other-Clerical Error | 3 | 0
Not completed — Other-Early termination | 6 | 10
Not completed — Other-Procedure | 1 | 1
Not completed — Other-Pregnancy | 2 | 4
Not completed — Other-Protocol Violation | 1 | 3
Not completed — Other-Lack of Efficacy | 1 | 0
Not completed — Other-Non Compliance | 2 | 0
Not completed — Other-Physician Decision | 1 | 1
Not completed — Other-Sponsor Decision | 10 | 12
Not completed — Other-Study Termination | 0 | 1
Not completed — Other-Study Withdrawn | 1 | 1
Not completed — Other-Site Stopped Communicating | 2 | 0
Not completed — Other-Lost to Follow-up | 1 | 0
Not completed — Other-Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Received Ferumoxytol in IDA-303: Participants received ferumoxytol or placebo during AMAG-FER-IDA-301 [NCT01114139]. Participants in AMAG-FER-IDA-303 who were found to have persistent or recurrent IDA, defined as hemoglobin <11.0 g/dL and TSAT <20% at any monthly evaluation visit, (with the exception of the Study Termination visit), began a 5-week TP and received a total of 2 doses of ferumoxytol 510 mg IV. The first IV 510 mg dose was administered on TP Day 1 (baseline) and second dose 2 to 8 (5±3) days after Dose 1, for a total cumulative dose of 1.02 g.
- Total: Total of all reporting groups
Arm/Group | Received Ferumoxytol in IDA-303 | Did Not Receive Ferumoxytol in IDA-303 | Total
Number analyzed (Participants) | 337 | 297 | 634
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.33) | 43.8 (13.26) | 44.9 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 269 | 573
  Male | 33 | 28 | 61

OUTCOME MEASURES:

1. Primary Outcome: Mean Change In Hemoglobin From TP Baseline To TP Week 5 Following The First Course Of Ferumoxytol
Description: Mean change in hemoglobin from TP Baseline (Day 1) to TP Week 5 following the first dose of ferumoxytol was calculated as: Hemoglobin Change = Hemoglobin (TP Week 5) - Hemoglobin (TP Baseline) TP Baseline was the most recent value measured on/after the screening or the closest monthly evaluation visit prior to Day 1 dosing of Course 1.
  Change from Baseline used an imputed value of 0 for missing values at the post-baseline visit.
Time Frame: TP Baseline (Day 1), TP Week 5
Population: ITT Population: Participants who received at least 1 dose of ferumoxytol and had evaluable data for hemoglobin at TP Baseline and TP Week 5 in AMAG-FER-IDA-303.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Ferumoxytol: Participants enrolled in AMAG-FER-IDA-303 who were found to have persistent or recurrent IDA, defined as hemoglobin <11.0 g/dL and TSAT <20% at any monthly evaluation visit, (with the exception of the Study Termination visit), began a 5-week TP and received a total of 2 doses of ferumoxytol 510 mg IV. The first IV 510 mg dose was administered on TP Day 1 (baseline) and second dose 2 to 8 (5±3) days after Dose 1, for a total cumulative dose of 1.02 g.
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 151
g/dL | 2.6 (1.55)
Statistical Analysis 1: Comparison: Ferumoxytol; Test type: Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Mean Change In Hemoglobin Following Each Course Of Ferumoxytol From TP Baseline To TP Week 5 Following Each Course Of Ferumoxytol After The First Course
Description: Mean change in hemoglobin from TP Baseline to TP Week 5 following each course of ferumoxytol after the first course was calculated for each participant as:
  Hemoglobin Change = Hemoglobin (TP Week 5) - Hemoglobin (TP Baseline) The first course of treatment with ferumoxytol for participants who had previously received placebo in AMAG-FER-IDA-301 was considered Course 1. The first course of treatment with ferumoxytol for participants who had previously received ferumoxytol in AMAG-FER-IDA-301 was considered Course 2; subsequent treatment courses were serially numbered.
Time Frame: TP Baseline (Day 1), TP Week 5 for Courses 1, 2, and 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 337
g/dL
  Course 1: number analyzed (Participants) | 151
  Course 1 | 2.6 (1.55)
  Course 2: number analyzed (Participants) | 244
  Course 2 | 1.5 (1.28)
  Course 3: number analyzed (Participants) | 69
  Course 3 | 1.1 (1.30)

3. Secondary Outcome: Percentage Of Participants With An Increase In Hemoglobin ≥2.0 g/dL At Any Time From TP Baseline To TP Week 5
Description: Proportion of participants with an increase in hemoglobin ≥2.0 g/dL at any time from TP Baseline to TP Week 5 following each course of ferumoxytol. The first course of treatment with ferumoxytol for participants who had previously received placebo in AMAG-FER-IDA-301 was considered Course 1. The first course of treatment with ferumoxytol for participants who had previously received ferumoxytol in AMAG-FER-IDA-301 was considered Course 2; subsequent treatment courses were serially numbered.
Time Frame: TP Baseline (Day 1), TP Week 5 for Courses 1, 2, and 3
Population: ITT Population: Participants who received at least 1 dose of ferumoxytol and had evaluable data for hemoglobin at TP Baseline and TP Week 5 in AMAG-FER-IDA-303.
  Participants with no post-baseline hemoglobin values were classified as not achieving the increase.
  Percentages are based on the number of participants in each course.
Measure: Number; unit: percentage of participants
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 337
percentage of participants
  Course 1: number analyzed (Participants) | 151
  Course 1 | 78.8
  Course 2: number analyzed (Participants) | 244
  Course 2 | 43.9
  Course 3: number analyzed (Participants) | 69
  Course 3 | 37.7

4. Secondary Outcome: Percentage Of Participants Who Achieved A Hemoglobin Level ≥12.0 g/dL At Any Time From TP Baseline To TP Week 5 Following Each Course Of Ferumoxytol
Description: Proportion of participants who achieved a hemoglobin level ≥12.0 g/dL at any time from TP Baseline to TP Week 5 following each course of ferumoxytol. The first course of treatment with ferumoxytol for participants who had previously received placebo in AMAG-FER-IDA-301 was considered Course 1. The first course of treatment with ferumoxytol for participants who had previously received ferumoxytol in AMAG-FER-IDA-301 was considered Course 2; subsequent treatment courses were serially numbered.
Time Frame: TP Baseline (Day 1), TP Week 5 for Courses 1, 2, and 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 337
percentage of participants
  Course 1: number analyzed (Participants) | 151
  Course 1 | 38.4
  Course 2: number analyzed (Participants) | 244
  Course 2 | 57.0
  Course 3: number analyzed (Participants) | 69
  Course 3 | 40.6

5. Secondary Outcome: Mean Change In TSAT Following Each Course Of Ferumoxytol From TP Baseline To TP Week 5 Following Each Course Of Ferumoxytol
Description: Mean change in TSAT from TP Baseline to TP Week 5 following each course of ferumoxytol.
Time Frame: TP Baseline (Day 1), TP Week 5 for Courses 1, 2, and 3
Population: ITT Population: Participants who received at least 1 dose of ferumoxytol and had evaluable data for TSAT at TP Baseline and TP Week 5 in AMAG-FER-IDA-303.
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 337
percentage of saturation
  Course 1: number analyzed (Participants) | 151
  Course 1 | 12.8 (10.19)
  Course 2: number analyzed (Participants) | 244
  Course 2 | 11.7 (12.47)
  Course 3: number analyzed (Participants) | 69
  Course 3 | 7.5 (9.13)

6. Secondary Outcome: Patient-reported Outcome Measure: Mean Change In Functional Assessment Of Chronic Illness Therapy (FACIT)-Fatigue Questionnaire From TP Baseline To TP Week 5 Following Each Course Of Ferumoxytol
Description: The FACIT-Fatigue questionnaire is a 13-item questionnaire designed and validated to specifically assess the presence and impact of treatment on fatigue and related symptoms, such as tiredness, on health-related quality of life in anemic participants with cancer. The questionnaire has 13 items, each measured on a 4-point Likert scale. Scoring ranges from 0 (the most fatigued) to 52 (the least fatigued) points, with higher scores representing better functioning or less fatigue.
  Mean change in FACIT-Fatigue questionnaire from TP Baseline to TP Week 5 following each course of ferumoxytol was calculated as:
  FACIT-Fatigue Score Change = FACIT-Fatigue Score (Week 5) - FACIT-Fatigue Score (Baseline).
  TP Baseline was the most recent value measured on/after the screening or the closest monthly evaluation visit prior to Day 1 dosing in each course.
  If the TP Week 5 FACIT-Fatigue Score value was missing, the change from TP Baseline was conservatively imputed as zero.
Time Frame: TP Baseline (Day 1), TP Week 5 for Courses 1, 2, and 3
Population: ITT Population: Participants who received at least 1 dose of ferumoxytol and had evaluable FACIT-Fatigue Questionnaire data at TP Baseline and TP Week 5 in AMAG-FER-IDA-303.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 337
units on a scale
  Course 1: number analyzed (Participants) | 151
  Course 1 | 6.9 (9.57)
  Course 2: number analyzed (Participants) | 244
  Course 2 | 4.1 (8.58)
  Course 3: number analyzed (Participants) | 69
  Course 3 | 1.5 (6.87)

7. Secondary Outcome: Time To Hemoglobin Increase Of ≥2.0 g/dL Or To A Hemoglobin Level Of ≥12.0 g/dL From Baseline
Description: Days to event was defined as the days from Baseline to the first time the participant met the criteria. Participants without any post-Baseline study visits were not included in this analysis.
  The first course of treatment with ferumoxytol for participants who had previously received placebo in AMAG-FER-IDA-301 was considered Course 1. The first course of treatment with ferumoxytol for participants who had previously received ferumoxytol in AMAG-FER-IDA-301 was considered Course 2; subsequent treatment courses were serially numbered.
Time Frame: TP Baseline (Day 1) up to TP Week 5 for Courses 1, 2, and 3
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 337
days
  Course 1: number analyzed (Participants) | 151
  Course 1 | 27.8 [22.0 to 36.0]
  Course 2: number analyzed (Participants) | 244
  Course 2 | 30.6 [22.0 to 37.0]
  Course 3: number analyzed (Participants) | 69
  Course 3 | 30.7 [22.0 to NA] — Insufficient number of participants with events.

ADVERSE EVENTS:
Description: The analysis of adverse events focused on treatment-emergent adverse events (TEAEs). A TEAE was defined as an event with an onset date and time on or after the first dosing start date and time, or on or after the first dosing start date if the onset time was missing. Thus, TEAEs by definition were only assessed in participants who received ferumoxytol in this extension study. Participants who did not receive ferumoxytol were not included the analysis of adverse events.
Groups:
- Received Ferumoxytol: Participants received ferumoxytol during AMAG-FER-IDA-301 [NCT01114139]. Participants enrolled in AMAG-FER-IDA-303 who were found to have persistent or recurrent IDA, defined as hemoglobin <11.0 g/dL and TSAT <20% at any monthly evaluation visit, (with the exception of the Study Termination visit), began a 5-week TP and received a total of 2 doses of ferumoxytol 510 mg IV. The first IV 510 mg dose was administered on TP Day 1 (baseline) and second dose 2 to 8 (5±3) days after Dose 1, for a total cumulative dose of 1.02 g.
Arm/Group | Received Ferumoxytol
Serious Adverse Events (participants affected / at risk) | 22/337
Other Adverse Events (participants affected / at risk) | 93/337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Received Ferumoxytol (N=337)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Received Ferumoxytol (N=337)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 17 (20)
Vomiting (Gastrointestinal disorders) | 10 (12)
Fatigue (General disorders) | 9 (9)
Oedema peripheral (General disorders) | 6 (6)
Pyrexia (General disorders) | 5 (5)
Nasopharyngitis (Infections and infestations) | 10 (10)
Sinusitis (Infections and infestations) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 19 (20)
Fall (Injury, poisoning and procedural complications) | 4 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Dizziness (Nervous system disorders) | 11 (11)
Headache (Nervous system disorders) | 24 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypertension (Vascular disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data have been received by Sponsor, the Site, and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 180 days to allow Sponsor to protect its interests.